CLINICAL TRIAL: NCT06400199
Title: Succesfull Fertility Preservation for Transfeminine Adolescents Via Semen Cryopreservation or Testicular Sperm Extraction
Brief Title: Fertility Preservation for Transfeminine Adolescents Via Semen Cryopreservation or Testicular Sperm Extraction
Acronym: TESE
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, J.A.F. Huirne, Prof. dr. J.A.F. Huirne, Amsterdam UMC, location VUmc
Other Study IDs: 2022.0303
Record Dates: First submitted 2023-11-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Gender Dysphoria, Adolescent
Keywords: Testicular sperm extraction; Fertility preservation; Puberty suppresion
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cohort study is to identify and predict parameters for successful testicular sperm extraction (TESE) procedures or semen cryopreservation more accurately and to evaluate the decision making process and the experience of postponing or temporarily discontinuing puberty suppression to undergo successful fertility preservation. in transfeminine (assigned male at birth) adolescents. The main question[s] it aims to answer are:

* What is the optimal timing for fertility preservation before the start or after temporarily discontinuing puberty suppression puberty suppression
* How do transfeminine adolescents and their parents experience the decision making process of fertility preservation
* how do transfeminine adolescents and their parents experienced postponing or temporarily discontinuing puberty suppression to undergo successful fertility preservation?

Participants will be asked to use their medical data, answer a questionnaire or participate in a (online) interview.

ELIGIBILITY:
Inclusion Criteria:

* Before start of puberty suppresion with a wish for fertility preservation
* After discontinuing puberty suppersion before the start of hormone therapy

Exclusion Criteria:

* Tanner stage > 4/5

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — assigned male at birth with a gender diverse gender identity
Study Population: assigned male at birth adolescents with gender dysphoria who wish fertilty preservation before the start of puberty suppression.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
What parameter is best in predicting successful fertility preservation (i.e. spermatazoa are present) | Most recent before the TESE of semen cryopreservation no longer than 3 months old
  Testicular volume
What parameter is best in predicting successful fertility preservation (i.e. spermatazoa are present) | Most recent before the TESE of semen cryopreservation no longer than 3 months old
  serum testosteron
What parameter is best in predicting successful fertility preservation (i.e. spermatazoa are present) | Most recent before the TESE of semen cryopreservation no longer than 3 months old
  serum LH
What parameter is best in predicting successful fertility preservation (i.e. spermatazoa are present) | Most recent before the TESE of semen cryopreservation no longer than 3 months old
  Serum FSH
What parameter is best in predicting successful fertility preservation (i.e. spermatazoa are present) | Most recent before the TESE of semen cryopreservation no longer than 3 months old
  Serum SHBG

SECONDARY OUTCOMES:
How do adolescents and parents experience fertility preservation | After refferal to fertility preservation specialist, after every 3 months after the start of Tanner 2, 1 month after the fertility preservation.
  self-constructed questionnaires and semi-structed interviews
How do adolescents and parents experience fertility preservation | 1 month post fertility preservation
  semi-structed interviews

CONTACTS AND LOCATIONS:
Overall Officials: Judith Huirne, MD, PHD, PROF, Principal Investigator — Amsterdam UMC
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, location AMC, Amsterdam
  - Amsterdam UMC, Location VU Medical Center, Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peri A, Ahler A, Gook D, O'Connell MA, Bourne H, Nightingale M, Telfer M, Jayasinghe Y, Pang KC. Predicting successful sperm retrieval in transfeminine adolescents after testicular biopsy. J Assist Reprod Genet. 2021 Oct;38(10):2735-2743. doi: 10.1007/s10815-021-02293-z. Epub 2021 Aug 23. PMID 34424432

DOCUMENTS (1):
  • Study Protocol (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT06400199/Prot_000.pdf